CLINICAL TRIAL: NCT01411917
Title: Transversus Abdominis Plane Blocks for Ileostomy Takedown: A Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Difficulties due to some factors
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-0249
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Ileostomy - Stoma
Keywords: surgical stomas; Nerve block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block group (Experimental): Patients in this group will have a preoperative, ultrasound guided injection of 30ml of 0.375% bupivacaine into the muscle plane between the transversus abdominis muscle and internal oblique muscles.
  Interventions: Procedure: Transversus abdominis plane block
- Placebo (Placebo Comparator): Patients in this group will have an ultrasound guided subcutaneous injection of 30 ml of sterile preservative free saline.
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — Ultrasound guidance will be utilized to inject 30ml of 0.375% bupivacaine into the muscular plane between the internal oblique and transversus abdominis muscles.

SUMMARY:
Consenting subjects will be randomized to receive injection of bupivacaine or placebo before surgery for ileostomy takedown (injection administered after general anesthesia has been administered). Pain and side effects will be assessed periodically after surgery using the verbal Numeric Rating pain Scores, including at the timepoint of 24 hours after surgery. All subjects in this study will be given toradol to ensure adequate pain control.

DETAILED DESCRIPTION:
Subject Enrollment

The charts of patients who are scheduled for ileostomy takedown surgery will be screened for eligibility the day before surgery by an investigator on this study. On the day of surgery, patients will be seen in their pre-operative holding area by a member of their anesthesia team or the acute pain team. They will be screened for eligibility for anesthesia and surgery. Once they are cleared for the operating room they will be seen by a resident, fellow, or attending for the acute pain service, who is an investigator on this study, to confirm eligibility for this study. A peripheral intravenous line will also be placed as is standard for the operating room. If it has been determined that they meet eligibility criteria they will have further discussion with the clinical trials coordinator or an investigator to determine if the patient would like to participate in this study. If they would like to proceed as a subject in this study they will be consented. The consent process will take place in a semi-enclosed space used in preoperative holding to consent for surgical procedures and anesthesia. Study investigators or coordinators will conduct the consent process.

Conduct of Study

Study Procedure Overview

The nurses will check the patient into the preoperative holding area and collect usual preoperative information. Once the patient has consented to be a part of this study they will be brought to the block room. Standard monitors will be placed and a time- out procedure will be performed, as is standard for all procedures which take place in the block room. Side of procedure will be verified. At this time the subject will be randomized to receive TAP block or placebo by random computer generated assignment that is in a sealed envelope. The study solution will be prepared by the regional anesthesiologist performing the procedure. The subject will receive sedation with midazolam and versed titrated to effect as is standard for all block placements. The subjects' abdomen on the side ipsilateral to the ileostomy will be sterilely prepared. The ultrasound will have a sterile dressing placed over the probe and a standard 21 gauge or 22 gauge b-bevel, 10 cm block needle will be flushed with the study solution. A syringe of 1% lidocaine will also be prepared to anesthetize the skin prior to insertion of the block needle. The ultrasound will be placed on the abdomen. Once a good view of the 3 muscle layers of interest is visualized (internal oblique, external oblique and transverses abdominis) the probe will be held still and the 1% lidocaine will be used to numb the skin. The block needle will be placed "in line" with the probe so that the entirety of the needle may be visualized during the procedure.

Treatment Study Procedure

The TAP block will be placed using a standardized ultrasound guided approach. Subjects assigned to the study group will have an injection of 30ml of 0.375% bupivacaine, a local anesthetic with 3mcg/ml of epinephrine placed into the plane between the internal oblique and the transversus abdominis. The needle will be aspirated every 5 ml to monitor for possible intravascular injection. During the injection the pulse and EKG will be monitored as well to screen for intravascular injection. Once the solution has been injected the needle will be removed from the skin and the area cleaned off with a dry cloth.

Control Study Procedure

The placebo block will be an ultrasound guided subcutaneous injection into the plane of tissue right before external oblique. The standard ultrasound guided approach will be used. The solution injected will be 30 ml of sterile preservative free saline. The reason we will choose to do this injection subcutaneously is because it will minimize patient risk from this injection. Subcutaneous injections will be far from the peritoneal cavity. By using normal saline for this injection we eliminate the very small risk of local anesthetic toxicity. Note that every subject, regardless of group assignment, will receive a very aggressive pain control regimen (IV PCA-patient controlled analgesia, toradol, scheduled tylenol, local wound infiltration) for adequate analgesia. Toradol is not routinely used and is added for purposes of aggressive pain control for all subjects in this study.

Follow up

Subjects will receive a general anesthetic for their surgical procedure. An appropriate dose of propofol will be used for induction of anesthesia. Fentanyl will be administered for intra-operative analgesia as deemed necessary by the anesthesia team caring for the patient in the operating room. No long acting opioids, ketamine, or local anesthetic infusions will be administered during the case. Dexamethasone (4 mg IV) will be administered at induction and zofran (4 mg IV) will be administered prior to emergence. Local infiltration of the wound with local anesthetic will be performed on all subjects, as is standard for this surgery. The local anesthetic used will be per surgeon preference.

After the Surgery

* All subjects will be started on a hydromorphone patient controlled analgesia (PCA) as well as toradol (15 mg IV q 6 hours for 24 hours).
* A member of the study protocol or the anesthesia acute pain service will evaluate all subjects in the PACU.

  * They will assess Numeric Rating pain Scores (NRS) 0-10 where 0 represents no pain and 10 represents the worst pain imaginable, vital signs, and the presence of side effects including nausea, vomiting and/or pruritis. This pain assessment is standard care and would happen regardless of study participation.

Day 2 (post operative day 1(POD1))

* Study personnel will evaluate all subjects the morning after surgery. They will assess current pain scores, duration of block (when known), and the presence of side effects including nausea, vomiting and/or pruritis. The assessment of pain scores will be the same assessment as is done on the day of surgery, but at the 24-hour post-surgery timepoint it is done by the study coordinator for research purposes.
* Medical records will be reviewed in order to collect information about subject's pain overnight and medication administration. We will also collect age, sex, height, weight, opioid usage (weekly, monthly, rarely), baseline pain score, and ASA physical status from the medical record.

Data Recording

After blocks are performed a procedure note will be entered into the medical record of the subject. The procedure note will document that the subject is enrolled in this study and that they may have received a TAP block with 30 ml of 0.375% bupivacaine with epinephrine. It will say that they also may have received a subcutaneous injection of normal saline. The note will document any complications encountered during block placement and the subjects' disposition at the time of completion of the block. A record of which subject has received what type of block, and solution, will be kept in a document held in a locked cabinet in the block room (within the operating room). This can be referenced and reported to the anesthesia team caring for the patient if issues arise during patient care which would necessitate unblinding. Otherwise, on post-operative day 1 (POD1), a procedure note documenting the actual procedure will be entered into the subject's medical chart. This will be done after the study data has been collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having an ileostomy takedown alone, on one side of abdomen
2. Ages 18-80 inclusive
3. English speaking
4. BMI less than 40
5. Ability to understand verbal pain scale
6. American Society of Anesthesiologists (ASA) Physical Status 1-3

Exclusion Criteria:

1. Allergy to local anesthetics
2. History of recent/current local or generalized infection
3. Immunocompromised
4. Significant psychiatric disease
5. History of opioid dependence
6. Pregnancy or lactation
7. A prisoner.
8. Significant liver disease
9. Contraindication to ondansetron or dexamethasone
10. Clinically significant cardiac or pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-08; Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Result] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Result] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block Group | Placebo
Started | 32 | 37
Completed | 32 | 36
Not Completed | 0 | 1
Not completed — Patient did not undergo scheduled surger | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block Group | Placebo | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.2) | 39.4 (13.5) | 38.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 19 | 24 | 43
Body Mass Index (BMI) kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 25.3 (4.3) | 25.1 (4.1) | 25.2 (4.2)
American Society of Anesthesiologists Physical Status Score (I-VI based on Health of Patient) [Median (Full Range); unit: units on a scale] — ASA I- A normal healthy patient. ASA II- A patient with mild systemic disease. ASA III- A patient with severe systemic disease. ASA IV- A patient with severe systemic disease that is a constant threat to life.
  ASA V- A moribund patient who is not expected to survive without the operation. ASA VI- A declared brain-dead patient whose organs are being removed for donor purposes.
  units on a scale | 2 [1 to 2] | 2 [1 to 2] | 2 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Postoperative Opioid Consumption
Description: We aim to evaluate whether patients consume less opioids, over the first 24 hours post-operatively following ileostomy takedown, with the addition of a pre-operative Transversus Abdominis Plane (TAP) block for analgesia.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 30 | 35
mg | 57.7 (49.3) | 77.8 (46.8)

2. Secondary Outcome: Pain Scores at Post-anesthesia Care Unit (PACU) Discharge
Description: 0-10 Pain Scale Numerical Rating Pain Scale. 0 represents no pain and 10 represents the worst pain imaginable.
Time Frame: Surgical PACU (Approximately 2 hours post-anesthesia)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 32 | 36
units on a scale | 3.3 (1.8) | 3.8 (2)

3. Secondary Outcome: Pain Scores at 24 Hours Post-block
Description: 0-10 Pain Scale Numerical Rating Pain Scale. 0 represents no pain and 10 represents the worst pain imaginable.
Time Frame: 24 hours post-block
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 30 | 35
units on a scale | 3.1 (2) | 2.5 (1.9)

4. Secondary Outcome: Time From PACU Recovery Room Admission Until Meeting Recovery Room Discharge Criteria
Time Frame: Approximately two hours post-anesthesia
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 32 | 36
Minutes | 29 (56.4) | 18 (37.4)

5. Secondary Outcome: Intra-operative Opioid Use
Description: Morphine Equivalents
Time Frame: Approximately 2-3 hours after block/placebo placement
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 32 | 36
mg | 31.1 (14.1) | 28.6 (8.9)

6. Secondary Outcome: PACU Opioid Use
Description: Morphine Equivalents
Time Frame: Approximately two hours post-anesthesia
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 32 | 36
mg | 8.8 (7.6) | 12.9 (9.9)

7. Secondary Outcome: Incidence of Post-operative Nausea
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 30 | 35
Participants | 10 | 14

8. Secondary Outcome: Time to Hospital Discharge
Description: This outcome is intended to assess the impact of the regional anesthesia technique on the amount of time that patients stayed in the hospital following their surgical procedure. This outcome is measured in hours.
Time Frame: Hours that patient spends in the hospital for their surgical procedure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAP Block Group | Placebo
Number analyzed (Participants) | 30 | 35
hours | 107.4 (58.4) | 97.6 (60.4)

ADVERSE EVENTS:
Arm/Group | TAP Block Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/36
Other Adverse Events (participants affected / at risk) | 0/32 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAP Block Group (N=32) | Placebo (N=36)
Postoperative Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes